CLINICAL TRIAL: NCT02760524
Title: Desensitizing Distressing Recollections in Cancer Patients
Acronym: NET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09D.182; JT 1487 (Other: JeffTrial Number)
Record Dates: First submitted 2015-09-29; First posted 2016-05-03 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Subjects will receive NET intervention treatment immediately
  Interventions: Behavioral: NET Intervention
- Control (Active Comparator): Subjects will receive NET intervention treatment and serve as a wait-list control
  Interventions: Behavioral: NET Intervention

INTERVENTIONS:
Behavioral: NET Intervention — Neuro-emotional Technique

SUMMARY:
The major goal of this study is to determine whether Neuro-Emotional Technique is a viable treatment option for decreasing distress in cancer patients. The potential advantages of NET are: 1) it is designed specifically to address distressing stimuli and unresolved emotional memories; 2) it is a brief, time-limited intervention; and 3) its multi-modal design may appeal to and benefit a broader range of patients than a single mode intervention

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* Distressing cancer-related recollection that has persisted for at least six months
* Distressing cancer-related recollection that causes physiological reactivity (i.e., increased heart rate and/or increased skin conductance level - SCL), as described in section 4.2.3.
* Received a cancer diagnosis at least 6 months prior to being contacted for participation in this study

Exclusion Criteria:

* Any current Major Mental Disorder, as assessed by Structured Clinical Interview for DSM IV Axis I Disorders (SCID - Clinical Version, First et al, 1997)
* History of Post-traumatic Stress Disorder
* Current active mood primary disorder prior to the cancer diagnosis (as per PI or designate)
* History or current diagnosis of substance or alcohol abuse or dependence (as per PI or designate)
* Use of psychotropic medications within the past month or current use of medications that would interfere with autonomic nervous system measures (benzodiazepines, barbiturates, major tranquilizers).
* Use of some psychotropic medications are allowed such as SSRIs and certain sleep aids, but dosages must be stable from six weeks prior to enrollment and throughout study period
* Any psychological or musculoskeletal problems that would interfere with psychophysiological assessments and treatment
* Currently receiving chemotherapy or radiation
* Are in the terminal stages of illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-04-11 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Post traumatic Cognitions Inventory | baseline/ 4 weeks/6 months follow up
  change from baseline Post Traumatic Cognitions Inventory score
State Trait Anxiety Inventory | baseline/4 weeks/6 months follow up
  change from baseline State Trait Anxiety Inventory score
Brief Symptom Inventory | baseline/4 weeks/6 month follow up
  change from baseline Brief Symptom Inventory

SECONDARY OUTCOMES:
Autonomal response to distressing recollections | baseline/4 weeks follow up
  change from baseline in autonomal response to distressing recollections
Genomic testing | baseline/ 4 weeks follow up
  change from baseline genomic testing before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Monti, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/